CLINICAL TRIAL: NCT02766127
Title: A Comparative Study of a Self-adhering Material in Dental Hypersensitivity in Xerostomic Patients Due to Radiotherapy
Brief Title: Effect of a Self-adhering Material in Dental Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Egle Milia, Prof, Università degli Studi di Sassari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000/CE
Record Dates: First submitted 2016-04-21; First posted 2016-05-09 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Dentin Sensitivity; Xerostomia
Keywords: radiotherapy
MeSH Terms: conditions — Dentin Sensitivity; Xerostomia | interventions — universal dentin sealant; Clearfil Protect Bond

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Xerostomic Patients (Experimental): Patients with evident clinical signs of xerostomia who experienced dentinal hypersensitivity after undergoing radiation therapy due to head and neck cancer.
  The following dental materials will be used following the manufacturers' instructions: Veritise Flow; Universal Dentin Sealant; Clearfil Protect Bond, and Flor-Opal® Varnish. In view of the treatment with the desensitizing agents, teeth were randomly assigned into four groups.
  the application of the materials will be made only once. The effectiveness will be evaluated: immediately after application and after 1, 4, 12 weeks.
  Interventions: Other: Veritise Flow; Other: Universal Dentin Sealant; Other: Clearfil Protect Bond; Other: Flor-Opal® Varnish

INTERVENTIONS:
Other: Veritise Flow — Self-adhering composite
  Other Names: Kerr Corporation, USA; Batch no. 3391829
Other: Universal Dentin Sealant — non-polymerizable, high molecular weight resin sealant
  Other Names: Ultradent Products Inc., USA; Batch no. 052809
Other: Clearfil Protect Bond — methacrylate-based resin, self-etching adhesive system
  Other Names: Kuraray Noritake Dental, Japan; Batch no. 041212
Other: Flor-Opal® Varnish — fluoride-based varnish
  Other Names: Ultradent Products Inc., USA; Batch no. 122005

SUMMARY:
Aim: To compare the desensitizing capacity of Vertise Flow™ (VF), a new self adhering material, in the treatment of dentine hypersensitivity (DH) in patients who are xerostomic due to radiotherapy for head and neck cancer.

Methods: A total of 17 patients were selected for the study. The study was conducted as a split-mouth randomized clinical trial comparing: 1) VF 2) Universal Dentin Sealant (UDS), 3) Clearfil Protect Bond (CPB) and 4) Flor-Opal® Varnish (FOV). Basal and stimulated salivary flow was recorded for each patient according to the method described by Sreebny. The pain experience was generated by a cold stimulus directly to a sensitive tooth surface and assessed using the Visual Analogue Scale (VAS). The response was recorded before the application of the materials (PRE-1), immediately after (POST-1), at 1-week (POST-2), 4-weeks (POST-3) and 12-week controls (POST-4).

DETAILED DESCRIPTION:
Participants The study was designed as a split-mouth randomized clinical trial. The protocol and informed consent forms were approved by the ethics committee at the University of Sassari (n° 1000/CE).

To participate in the study, all the subjects were carefully informed about the study's purpose, risks and benefits.

The study inclusion criteria were the following:

* Generally good health despite the seriousness of their illness;
* A clinical reduction of salivary flow;
* The presence of two or three teeth which were hypersensitive to stimulation with a blast of air.

In addition, patients were considered suitable for the study if they had sensitive teeth showing abrasion, erosion or recession with the exposure of the cervical dentine.

The study exclusion criteria were:

* teeth with subjective or objective evidence of carious lesions, pulpitis, restorations, premature contact, cracked enamel, active periapical infection or that had received periodontal surgery or root-planning up to 6 months prior to the investigation;
* patients who had received professional desensitizing therapy during the previous 3 months;
* patients who had used desensitizing toothpaste in the last 6 weeks. Patients were also excluded if they were under significant medication that could have interfered with pain perception (e.g., antidepressants, anti-inflammatory drugs, sedatives, and muscle relaxants).

Clinical Procedure

Saliva collection

All salivary assessments were performed in the absence of acute sialadenitis. All assessments were performed by the same observer. The flow rate was determined in every person according to the method described by Sreebny. Saliva was collected in a standardised manner. Patients were instructed not to eat, drink, or smoke for 90 minutes before the sialometric assessment. All assessments were performed at a fixed time of the day, between 10 am and 1 pm, in order to minimise fluctuations related to a circadian rhythm of salivary secretion and composition. The whole saliva sample was collected in pre-weighed plastic tubes using electronic scales.

Unstimulated salivary secretions were collected for 5 min with the patient seated in an upright position, with the head tilted forward . When possible the tongue, cheek and lip movements were limited during the procedure. At the end of the collection period the patient had to expectorate saliva into the test-tube. Stimulated whole saliva samples were collected by asking patients to chew a small block of paraffin wax or chewing gum. All the saliva secreted for 5 min was then collected in the test-tube. Measuring vessels were weighed after each collection using an electronic scales, and salivary flow rate was expressed in ml/min, which is nearly equivalent to g/min (31). A secretion rate < 0.1-0.2 ml/min for unstimulated flow and < 0.5-0.7 ml/min for stimulated flow was considered as an objective sign of hyposalivation.

Assessment of hypersensitivity and application of desensitizing agents.

A week before the experiment, patients received oral prophylaxis. Non-fluoride toothpaste (Biorepair, Coswell), a soft toothbrush (Oral-B Sensitive Advantage, Procter & Gamble) and oral hygiene instructions were also provided. The level of sensitivity experienced by each patient was considered as independent of the position of the hypersensitive tooth in the oral cavity. The pain experience was assessed by a Visual Analogue Scale (VAS) using the methodology described in our previous study. The pain experience was measured using a VAS graded from 1 to 10. The pain stimulus was given by one examiner with the same equipment yielding similar air pressure each time, while another one performed the treatments. The same operator carried out the sensitivity test evaluating the subject's response before the application of the materials (PRE-1), immediately after (POST-1), after 1 week (POST-2), 4 weeks (POST-3), and 12 weeks (POST-4) .

The following dental materials were used following the manufacturers' instructions: Verities Flow™ (VF) (Kerr Corporation, Orange, CA, USA), a self-adhering composite; Universal Dentin Sealant (UDS) (Ultradent Products Inc., South Jordan, UT, USA), a biocompatible, non-polymerizable, high molecular weight resin sealant in alcohol solvent; Clearfil Protect Bond (CPB), (Kuraray Noritake Dental, Osaka, Japan) a methacrylate-based resin, self-etching adhesive system, and Flor-Opal® Varnish (FOV), (Ultradent Products Inc., South Jordan, UT, USA), a fluoride-based varnish.

In view of the treatment with the desensitizing agents, teeth were randomly assigned into four groups (N = per group).

ELIGIBILITY:
Inclusion Criteria:

* Generally good health despite the seriousness of their illness;
* A clinical reduction of salivary flow;
* The presence of two or three teeth which were hypersensitive to stimulation with a blast of air.

In addition, patients were considered suitable for the study if they had sensitive teeth showing abrasion, erosion or recession with the exposure of the cervical dentine.

Exclusion Criteria:

* teeth with subjective or objective evidence of carious lesions, pulpitis, restorations, premature contact, cracked enamel, active periapical infection or that had received periodontal surgery or root-planning up to 6 months prior to the investigation;
* patients who had received professional desensitizing therapy during the previous 3 months;
* patients who had used desensitizing toothpaste in the last 6 weeks. Patients were also excluded if they were under significant medication that could have interfered with pain perception (e.g., antidepressants, anti-inflammatory drugs, sedatives, and muscle relaxants).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of change of dentinal hypersensitivity after treatment | before the treatment (PRE-1), immediately after (POST-1), after 1 week (POST-2), 4 weeks (POST-3), and 12 weeks (POST-4).
  The pain experience was assessed by a Visual Analogue Scale (VAS) using the methodology. The VAS scale consisted of a horizontal line that was 100 mm long, on which 'no pain' was marked on the right-hand extremity and 'unbearable pain' on the other. The patients expressed the intensity of the pain experienced by placing a mark at any point along the continuum. The distance, expressed in millimetres, from the right edge of 'no pain' was used as the VAS score. Each patient was asked to rate the perception of discomfort after the application of air via a dental syringe at 45-60 psi, 1 cm at the cervical third of the tooth after removing supragingival plaque with a low- speed handpiece with pumice powder and without fluoride. The adjacent teeth were covered by cotton rolls. The stimulus was delivered until reaction or up to a maximum duration of 10 s by the same examiner with the same equipment yielding similar air pressure each time.

CONTACTS AND LOCATIONS:
Overall Officials: Egle Milia, Prof, Principal Investigator — Università degli Studi di Sassari
Locations (1):
- Complex Operative Unit of Dentistry, Sassari, Sassari, Italy

IPD SHARING:
Plan to Share IPD: No
Not a plan for data sharing has been established. But, for anyone researcher would like to have this information, simply they may request them to us directly.

REFERENCES:
- [Background] Pinna R, Campus G, Cumbo E, Mura I, Milia E. Xerostomia induced by radiotherapy: an overview of the physiopathology, clinical evidence, and management of the oral damage. Ther Clin Risk Manag. 2015 Feb 4;11:171-88. doi: 10.2147/TCRM.S70652. eCollection 2015. PMID 25691810
- [Background] Pinna R, Bortone A, Sotgiu G, Dore S, Usai P, Milia E. Clinical evaluation of the efficacy of one self-adhesive composite in dental hypersensitivity. Clin Oral Investig. 2015 Sep;19(7):1663-72. doi: 10.1007/s00784-014-1390-3. Epub 2015 Jan 23. PMID 25609032
- [Background] Milia E, Castelli G, Bortone A, Sotgiu G, Manunta A, Pinna R, Gallina G. Short-term response of three resin-based materials as desensitizing agents under oral environmental exposure. Acta Odontol Scand. 2013 May-Jul;71(3-4):599-609. doi: 10.3109/00016357.2012.700063. Epub 2012 Aug 15. PMID 22891890